CLINICAL TRIAL: NCT07012174
Title: Body Mass Index and Lipid Metabolism in Relation to Anti-PD-1 Immunotherapy in Colorectal Cancer: A Retrospective Observational Study With Lipidomic Profiling
Brief Title: Impact of Body Mass Index and Lipid Metabolism on Anti-PD-1 Immunotherapy Outcomes in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Director of the Department of Colorectal Surgery, Sun Yat-sen University
Other Study IDs: No.G2023-176-01; 82373431, 82202947, 82473395, (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-05-28; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to evaluate the impact of body mass index (BMI) and dyslipidemia on the effectiveness of anti-PD-1 immunotherapy in patients with colorectal cancer (CRC). A total of 142 patients treated with immune checkpoint inhibitors at Sun Yat-sen University Cancer Center were retrospectively analyzed. The study assessed progression-free survival (PFS) based on BMI and lipid profiles. Lipidomic profiling was also performed to explore potential metabolic mechanisms. The aim of this study was to identify simple, clinically applicable biomarkers to guide treatment decisions for CRC patients receiving immunotherapy.

DETAILED DESCRIPTION:
This retrospective observational study investigates the prognostic value of body mass index (BMI) and dyslipidemia in colorectal cancer (CRC) patients treated with anti-PD-1 immune checkpoint inhibitors (ICIs). A total of 142 patients were included, all of whom received at least two cycles of PD-1 inhibitors, including Camrelizumab, Nivolumab, Pembrolizumab, Sintilimab, Tislelizumab, or Toripalimab, at Sun Yat-sen University Cancer Center between January 1, 2019, and December 31, 2022.

The primary objective of the study was to evaluate progression-free survival (PFS) stratified by BMI and lipid profile status. Patients were grouped by BMI into normal (<24 kg/m²) and overweight (≥24 kg/m²) categories, based on WHO standards for the Chinese population. Dyslipidemia was defined according to standard lipid thresholds. Kaplan-Meier and Cox proportional hazard models were used for survival analysis. Additionally, a subset of 12 patients underwent pre-treatment serum lipidomic profiling using ultra-performance liquid chromatography-tandem mass spectrometry (UPLC-MS/MS) to explore potential metabolic mechanisms contributing to differential responses.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years at time of diagnosis

Histologically confirmed colorectal adenocarcinoma

Received at least two doses of anti-PD-1 immune checkpoint inhibitor therapy (e.g., Camrelizumab, Nivolumab, Pembrolizumab, Sintilimab, Tislelizumab, or Toripalimab)

Availability of baseline body mass index (BMI) and lipid profile within 30 days prior to ICI initiation

Adequate clinical records for retrospective data collection

Signed informed consent for data usage (if applicable to retrospective cohort)

Exclusion Criteria:

Participation in another interventional clinical trial during the study period

Incomplete PD-1 treatment (< 2 cycles)

Severe immune-related adverse events leading to early discontinuation of immunotherapy

Missing or incomplete BMI or lipid profile data

Loss to follow-up prior to outcome assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) with histologically confirmed colorectal adenocarcinoma who received at least two cycles of anti-PD-1 immune checkpoint inhibitor therapy at Sun Yat-sen University Cancer Center between January 2019 and December 2022. All participants had available baseline BMI and lipid profile data. The cohort includes both males and females, with a mix of MSI-H and MSS cases, across various disease stages.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | Up to 36 months
  Time from initiation of anti-PD-1 therapy to documented disease progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Ding, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No